CLINICAL TRIAL: NCT03048006
Title: Evaluation of Dotarem Safety
Brief Title: Post-marketing Surveillance Study for Evaluation of Dotarem Safety
Status: Completed | Type: Observational
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: DGD-55-005
Record Dates: First submitted 2017-02-01; First posted 2017-02-09 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Contrast-enhanced MRI With Dotarem
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; gadoterate meglumine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All included patients: All included patients underwent MRI with Dotarem
  Interventions: Procedure: MRI with Dotarem

INTERVENTIONS:
Procedure: MRI with Dotarem
  Other Names: MRI with gadoteric acid/gadoterate meglumine

SUMMARY:
Guerbet conducted a non-interventional post-marketing surveillance study on its Magnetic Resonance Imaging (MRI) contrast agent Dotarem (gadoteric acid/gadoterate meglumine). The aim of this study, which was conducted in accordance with section 67, paragraph 6 of the German drug regulation, Arzneimittelgesetz, was to gain additional insights into the diagnostic efficacy, reliability and safety of Dotarem in routine practice using the most up-to-date MRI techniques and application methods.

DETAILED DESCRIPTION:
Diagnostic efficacy was assessed by the following endpoints: diagnostic value ("yes"/"no") and imaging quality (5-step scale from "excellent" to "very poor"). Safety was evaluated on the basis of the frequency and seriousness of adverse events that occurred following Dotarem injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine MRI using the MRI contrast medium Dotarem

Exclusion Criteria:

-

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients undergoing routine MRI using the MRI contrast medium Dotarem
Sampling Method: Non-Probability Sample
Enrollment: 44456 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Included Patients
Started | 44456
Completed | 44456
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Included Patients
Number analyzed (Participants) | 44456
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was missing for 167 patients.
  years
    number analyzed (Participants) | 44289
    (all) | 52.3 (16.9)
Age, Customized [Count of Participants; unit: Participants] — Population: Age was missing for 167 patients.
  Participants
    <2 years: number analyzed (Participants) | 44289
    <2 years | 1
    between 2 and 11 years: number analyzed (Participants) | 44289
    between 2 and 11 years | 81
    between 12 and 17 years: number analyzed (Participants) | 44289
    between 12 and 17 years | 617
    ≥18 years: number analyzed (Participants) | 44289
    ≥18 years | 43590
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender was missing for 687 patients.
  Participants
    number analyzed (Participants) | 43769
    Female | 24254
    Male | 19515
Risk factors [Count of Participants; unit: Participants] — Risk factors were recorded before the MRI examination Population: Out of the 44,456 patients, 11,006 showed at least one risk factor. Several risk factors could be reported for the same patient.
  Participants
    Known allergies | 6871
    History of a reaction to a contrast agent | 176
    Bronchial asthma | 630
    Beta-blocker treatment | 648
    Coronary heart disease | 824
    Heart failure | 413
    Hypertension | 2479
    Liver dysfunction | 121
    Central nervous system disorders | 560
    Other | 858

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events
Description: The frequency of adverse events (serious and non-serious) that occurred following injection of Dotarem was recorded.
Time Frame: From the beginning of the MRI procedure to 30-60 min after
Measure: Number; unit: adverse events
Arm/Group | All Included Patients
Number analyzed (Participants) | 44456
adverse events | 225

2. Secondary Outcome: Diagnostic Value
Description: Diagnostic value was evaluated by answering "yes" or "no" to the following question "Were you able to make a diagnosis based on the test results ?"
Time Frame: During MRI procedure
Population: Diagnostic value was missing for 77 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Patients
Number analyzed (Participants) | 44379
Participants
  Diagnosis achieved | 44312
  Diagnosis not achieved | 67

3. Secondary Outcome: Image Quality
Description: Image quality was evaluated with a 5-step scale from "excellent" to "very poor" ("excellent/very good"; "good"; "moderate"; "poor" and "very poor")
Time Frame: During MRI procedure
Population: Image quality was missing for 108 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Patients
Number analyzed (Participants) | 44348
Participants
  Excellent | 25580
  Good | 18218
  Moderate | 516
  Poor | 32
  Very Poor | 2

ADVERSE EVENTS:
Time Frame: From the beginning of the MRI procedure to 30-60 min after
Description: Several adverse events could be reported for the same patient.
Arm/Group | All Included Patients
All-Cause Mortality (participants affected / at risk) | 0/44456
Serious Adverse Events (participants affected / at risk) | 7/44456
Other Adverse Events (participants affected / at risk) | 132/44456
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Included Patients (N=44456)
Vomiting (Gastrointestinal disorders) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oral pruritus (Gastrointestinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Included Patients (N=44456)
Cardiovascular disorder (Cardiac disorders) | 6 (6)
Palpitations (Cardiac disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 69 (69)
Retching (Gastrointestinal disorders) | 5 (5)
Swollen tongue (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 21 (21)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Feeling hot (General disorders) | 3 (3)
Injection site erythema (General disorders) | 1 (1)
Injection site extravasation (General disorders) | 2 (2)
Injection site irritation (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 1 (1)
Local swelling (General disorders) | 2 (2)
Malaise (General disorders) | 5 (5)
Oedema mucosal (General disorders) | 1 (1)
Temperature intolerance (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2)
Contrast media allergy (Immune system disorders) | 1 (1)
Drug administration error (Injury, poisoning and procedural complications) | 2 (2)
Blood pressure decreased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 9 (9)
Dizziness postural (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (4)
Tremor (Nervous system disorders) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 11 (11)
Flushing (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pallor (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No